CLINICAL TRIAL: NCT02366910
Title: Dehydration of Omafilcon A Contact Lenses Versus Delefilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-45
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- omafilcon A (Experimental): Each subject will be randomized to wear the test lens in one eye and control lens in the other eye (contra lateral design).
  Interventions: Device: omafilcon A; Device: delefilcon A
- delefilcon A (Active Comparator): Each subject will be randomized to wear the test lens in one eye and control lens in the other eye (contra lateral design).
  Interventions: Device: omafilcon A; Device: delefilcon A

INTERVENTIONS:
Device: omafilcon A — Each subject randomized to wear either the test or control in either the left of right eye.
Device: delefilcon A — Each subject randomized to wear either the test or control in either the left of right eye.

SUMMARY:
The study will explore in vivo lens dehydration rates across a 12hr wear period for the study lenses.

DETAILED DESCRIPTION:
The study will explore in vivo lens dehydration rates across a 12hr wear period for the study lenses. The primary outcome variable for this study is the loss in lens weight over the day, which will indicate the amount of dehydration that has occured.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is a current wearer of soft contact lenses and has worn them (any brand) more than 3 months.
5. Is able to wear lenses for at least 12 hours a day.

Exclusion Criteria:

1. Is participating in any concurrent clinical study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Has undergone refractive error surgery;

   * *For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydon Jones, PhD FC, Principal Investigator — Director, Centre for Contact Lens Research; Farah Panjwani, BSc RAQ, Principal Investigator — Univerisy of Waterloo
Locations (1):
- University of Waterloo School of Optometry, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye (contra lateral design).
  omafilcon A: Each subject randomized to wear either the test or control in either the left of right eye.
  delefilcon A: Each subject randomized to wear either the test or control in either the left of right eye.
Period: Overall Study
Arm/Group | Overall Participants
Started | 26
Completed | 21
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Overall Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (10.1)
Age, Continuous [Median (Full Range); unit: years] | 24 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Water Content (Mean) of Omafilcon A and Delefilcon A
Description: Comparison between lens types up to and at 12 hours of wear for the absolute change in water content (WC).
Time Frame: 12 Hours of Wear
Population: Because of the outliers across three participants, the sample size for statistical analysis is reduced to 18 pairs.
Measure: Mean (Standard Deviation); unit: absolute WC change
Arm/Group | Omafilcon A | Delefilcon A
Number analyzed (Participants) | 18 | 18
absolute WC change | 1.59 (0.85) | 3.82 (1.75)

2. Primary Outcome: Absolute Change in Water Content (Median) of Omafilcon A and Delefilcon A
Description: Comparison between lens types up to and at 12 hours of wear for the absolute change in water content (WC).
Time Frame: 12 Hours of Wear
Population: Because of the outliers across three participants, the sample size for statistical analysis is reduced to 18 pairs.
Measure: Median (Full Range); unit: absolute WC change
Arm/Group | Omafilcon A | Delefilcon A
Number analyzed (Participants) | 18 | 18
absolute WC change | 1.20 [0.21 to 3.01] | 3.38 [0.37 to 7.25]

3. Primary Outcome: Moisture Retention (Mean) of Omafilcon A and Delefilcon A
Description: Comparison between lens types up to and at 12 hours of wear of moisture retention by measuring relative percentage dehydration (RPD).
Time Frame: 12 Hours
Population: Because of the outliers across three participants, the sample size for statistical analysis is reduced to 18 pairs.
Measure: Mean (Standard Deviation); unit: percentage of dehyrdation
Arm/Group | Omafilcon A | Delefilcon A
Number analyzed (Participants) | 18 | 18
percentage of dehyrdation | 2.58 (1.38) | 11.5 (5.2)

4. Primary Outcome: Moisture Retention (Median) of Omafilcon A and Delefilcon A
Description: as for outcome 3
Time Frame: 12 Hours
Population: Because of the outliers across three participants, the sample size for statistical analysis is reduced to 18 pairs.
Measure: Median (Full Range); unit: percentage of dehyrdation
Arm/Group | Omafilcon A | Delefilcon A
Number analyzed (Participants) | 18 | 18
percentage of dehyrdation | 1.98 [0.35 to 4.90] | 9.89 [1.18 to 21.44]

ADVERSE EVENTS:
Time Frame: From dispense up to 12 hour for each study lenses
Arm/Group | Omafilcon A | Delefilcon A
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.